CLINICAL TRIAL: NCT02088073
Title: Multicenter, Multi-phase, Multi-dose, Prospective, Double-blind, Placebo-controlled, Maintenance Study of Safety and Efficacy of ZS (Microporous, Fractionated, Protonated Zirconium Silicate) in Hyperkalemia.
Brief Title: Safety & Efficacy of Zirconium Silicate Dosed for 28 Days in Hyperkalemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ZS-004
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate; zircon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Sodium zirconium cyclosilicate 10 g three times daily (Experimental): Sodium zirconium cyclosilicate 10 g three times daily for 48 hours (acute phase)
  Interventions: Drug: Sodium zirconium cyclosilicate
- Placebo once daily (Placebo Comparator): Randomized to mimic doses of experimental drug administered once daily with breakfast for 28 days.
  Interventions: Drug: Placebo
- Sodium zirconium cyclosilicate 5 g once daily (Experimental): Sodium zirconium cyclosilicate (ZS) 5 g once daily for 28 days (maintenance phase)
  Interventions: Drug: Sodium zirconium cyclosilicate
- Sodium zirconium cyclosilicate 10 g once daily (Experimental): Sodium zirconium cyclosilicate (ZS) 10 g once daily for 28 days (maintenance phase)
  Interventions: Drug: Sodium zirconium cyclosilicate
- Sodium zirconium cyclosilicate 15 g once daily (Experimental): Sodium zirconium cyclosilicate (ZS) 15 g once daily for 28 days (maintenance phase)
  Interventions: Drug: Sodium zirconium cyclosilicate

INTERVENTIONS:
Drug: Sodium zirconium cyclosilicate — Sodium zirconium cyclosilicate
  Other Names: ZS; Microporous, Fractionated, Protonated Zirconium Silicate; Zirconium Silicate
  Arms: Sodium zirconium cyclosilicate 10 g once daily; Sodium zirconium cyclosilicate 10 g three times daily; Sodium zirconium cyclosilicate 15 g once daily; Sodium zirconium cyclosilicate 5 g once daily
Drug: Placebo — Randomized to mimic doses of experimental drug administered once daily with breakfast for 28 days (maintenance phase)
  Other Names: Silicilate microcrystaline cellulose
  Arms: Placebo once daily

SUMMARY:
It is hypothesized that ZS is more effective than placebo control (alternative hypothesis) in maintaining mean double-blind randomized maintenance phase (DBRMP) Day 8-29 serum potassium levels (3.5 - 5.0 mmol/l, inclusive) among hyperkalemic subjects in whom normokalemia was established during the open-label acute phase versus no difference between each ZS dose (highest to lowest) versus placebo control (null hypothesis).

DETAILED DESCRIPTION:
Approximately 275 subjects with hyperkalemia (two consecutive i-STAT potassium levels ≥ 5.1 mmol/l, taken 60 minutes apart at baseline) will be enrolled in the Open-label Acute Phase to provide 232 subjects in the Double Blind Randomized Maintenance Phase.

Initially all subjects will receive open-label ZS at a dose of 10g three times a day (tid) for 48 hours (AP). Subjects who achieve normokalemia (i-STAT potassium values between 3.5 to 5.0 mmol/l, inclusive) on the morning of Study Day 3 (after 6 doses of 10g ZS) will then, in a double-blind fashion, be randomized 4:4:4:7 to receive one of three doses of ZS (5g, 10g or 15g) or placebo control, qd for the following 28 days (DBRMP).

Safety and tolerability will be assessed on an ongoing basis by an Independent Data Monitoring Committee (iDMC). Each active dose group in the DBRMP will consist of 49 subjects and the placebo control group will consist of 85 subjects for a total of 232 subjects to detect a 0.6 effect size difference between each ZS dose (from highest to lowest) and placebo control; the 4:4:4:7 allocation optimizes the multiple comparisons to the placebo control for the DBRMP.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Over 18 years of age.
* Two consecutive i-STAT potassium values, measured 60-minutes apart, both ≥5.1 mmol/l and measured within 1 day of the first ZS dose on AP Study Day 1.
* Ability to have repeated blood draws or effective venous catheterization.
* Women of childbearing potential must be using two forms of medically acceptable contraception (at least one barrier method) and have a negative pregnancy test at AP Study Day 1. Women who are surgically sterile or those who are post-menopausal for at least 2 years are not considered to be of childbearing potential.

Exclusion Criteria:

* Pseudohyperkalemia signs and symptoms, such as excessive fist clenching hemolyzed blood specimen, history of severe leukocytosis or thrombocytosis.
* Subjects treated with lactulose, Xifaxan or other non-absorbed antibiotics for hyperammonemia within 7 days prior to the first dose of study drug.
* Subjects treated with resins (such as sevelamer acetate or sodium polystyrene sulfonate [SPS; e.g. Kayexalate®]), calcium acetate, calcium carbonate, or lanthanum carbonate, within 7 days prior to the first dose of study drug.
* Subjects with a life expectancy of less than 3 months.
* Subjects who are severely physically or mentally incapacitated and who in the opinion of investigator are unable to perform the subjects' tasks associated with the protocol.
* Women who are pregnant, lactating, or planning to become pregnant.
* Subjects with diabetic ketoacidosis.
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
* Known hypersensitivity or previous anaphylaxis to ZS or to components thereof.
* Randomization into the previous ZS-002 or ZS-003 studies.
* Treatment with a drug or device within the last 30 days that has not received regulatory approval at the time of study entry.
* Subjects with cardiac arrhythmias that require immediate treatment.
* Subjects on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2015-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Chair — ZS Pharma, Inc.
Locations (46):
- United States (38):
  - Anniston, Alabama
  - Huntsville, Alabama
  - Scottsboro, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - Hawaiian Gardens, California
  - Los Angeles, California
  - Paramount, California
  - Riverside, California
  - Atlantis, Florida
  - Bradenton, Florida
  - Brandon, Florida
  - Brooksville, Florida
  - DeLand, Florida
  - Edgewater, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Summerfield, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Columbus, Georgia
  - Decatur, Georgia
  - Evergreen Park, Illinois
  - Joliet, Illinois
  - Shreveport, Louisiana
  - Auburn, Maine
  - Chesterfield, Michigan
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Flushing, New York
  - Altoona, Pennsylvania
  - Providence, Rhode Island
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - Chattanooga, Tennessee
  - San Antonio, Texas
- Australia (5):
  - Gosford, New South Wales
  - Woolloongabba, Queensland
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria
- South Africa (3):
  - Meyerspark
  - Port Elizabeth
  - Somerset West

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430
- [Derived] Amin AN, Menoyo J, Singh B, Kim CS. Efficacy and safety of sodium zirconium cyclosilicate in patients with baseline serum potassium level >/= 5.5 mmol/L: pooled analysis from two phase 3 trials. BMC Nephrol. 2019 Dec 2;20(1):440. doi: 10.1186/s12882-019-1611-8. PMID 31791288
- [Derived] Kosiborod M, Rasmussen HS, Lavin P, Qunibi WY, Spinowitz B, Packham D, Roger SD, Yang A, Lerma E, Singh B. Effect of sodium zirconium cyclosilicate on potassium lowering for 28 days among outpatients with hyperkalemia: the HARMONIZE randomized clinical trial. JAMA. 2014 Dec 3;312(21):2223-33. doi: 10.1001/jama.2014.15688. PMID 25402495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 44 sites in the United States, Australia, and South Africa from 31 March 2014 to 08 August 2014
Pre-assignment Details: Subjects with hyperkalemia (i-STAT potassium value ≥ 5.1 mmol/L) were enrolled in the Acute Phase (AP) and were to be treated with ZS 10 g TID for the 48 hours.Subjects who achieved normokalemia during the AP were randomized to 1 of 3 doses of ZS (5 g, 10 g,or 15 g) or placebo for a further 28 days (Maintenance Phase [MP]).
Groups:
- ZS 10 g Three Times Daily (Acute Phase): Sodium zirconium cyclosilicate (ZS) 10 g, three times daily (TID), orally as a suspension for 48 hours.
- Placebo Comparator (Maintenance Phase): Placebo to mimic doses of experimental drug once daily between Days 8 to 29, inclusive.
- ZS 5 g Once Daily (Maintenance Phase): Sodium zirconium cyclosilicate (ZS) 5 g, once daily, orally as a suspension between Days 8 to 29, inclusive.
- ZS 10 g Once Daily (Maintenance Phase): Sodium zirconium cyclosilicate (ZS) 10 g, once daily, orally as a suspension between Days 8 to 29, inclusive.
- ZS 15 g Once Daily (Maintenance Phase): Sodium zirconium cyclosilicate (ZS) 15 g, once daily, orally as a suspension between Day 8 to 29, inclusive.
Period: Acute Phase
Arm/Group | ZS 10 g Three Times Daily (Acute Phase) | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Started | 258 | 0 | 0 | 0 | 0
Completed | 251 | 0 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0 | 0
Not completed — Hyperkalemia | 2 | 0 | 0 | 0 | 0
Period: Maintanance Phase
Arm/Group | ZS 10 g Three Times Daily (Acute Phase) | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Started | 0 | 85 | 45 | 51 | 56
Completed | 0 (251 subjects completed the AP; 240 were eligible to enter the MP. 237 entered the MP.) | 75 | 40 | 44 | 49
Not Completed | 0 | 10 | 5 | 7 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor's decision | 0 | 2 | 0 | 2 | 1
Not completed — Hypo- or hyperkalemia | 0 | 3 | 0 | 3 | 1
Not completed — Miscellaneous | 0 | 2 | 1 | 2 | 1
Not completed — Met ECG withdrawal criteria | 0 | 0 | 1 | 0 | 2
Not completed — Subject compliance | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Some participants contributed to more than one baseline group. 258 participants entered the acute phase; 251 completed the acute phase. Of these 251 participants, 240 were eligible for the maintenance phase. Three participants did not enter the maintenance phase; 237 participants were randomized for the maintenance phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | ZS 10 g Three Times Daily (Acute Phase) | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase) | Total
Number analyzed (Participants) | 258 | 85 | 45 | 51 | 56 | 495
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Acute Phase | 64.0 (12.72) | NA (NA) — This field does not apply to the Acute Phase of the study. | NA (NA) — This field does not apply to the Acute Phase of the study. | NA (NA) — This field does not apply to the Acute Phase of the study. | NA (NA) — This field does not apply to the Acute Phase of the study. | 64.0 (12.72)
  Maintenance Phase | NA (NA) — This field does not apply to the Maintenance Phase of the study. | 64.3 (12.13) | 61.5 (16.89) | 63.8 (9.97) | 64.9 (12.85) | 63.80 (13.01)
Sex/Gender, Customized [Number; unit: Participants]
  Female, Acute Phase | 109 | 0 | 0 | 0 | 0 | 109
  Male, Acute Phase | 149 | 0 | 0 | 0 | 0 | 149
  Female, Maintenance Phase | 0 | 41 | 18 | 24 | 16 | 99
  Male, Maintenance Phase | 0 | 44 | 27 | 27 | 40 | 138
Race/Ethnicity, Customized [Number; unit: Participants]
  White, Acute Phase | 215 | 0 | 0 | 0 | 0 | 215
  Black or African American, Acute Phase | 37 | 0 | 0 | 0 | 0 | 37
  Asian, Acute Phase | 5 | 0 | 0 | 0 | 0 | 5
  Native Hawaiian or other Pacific Islander, AP | 1 | 0 | 0 | 0 | 0 | 1
  Other, Acute Phase | 2 | 0 | 0 | 0 | 0 | 2
  Multiple Races indicated, Acute Phase | 1 | 0 | 0 | 0 | 0 | 1
  White, Maintenance Phase | 0 | 73 | 36 | 44 | 46 | 199
  Black or African American, Maintenance Phase | 0 | 10 | 8 | 5 | 9 | 32
  Asian, Maintenance Phase | 0 | 3 | 0 | 1 | 1 | 5
  Native Hawaiian or other Pacific Islander, MP | 0 | 1 | 0 | 0 | 0 | 1
  Other, Maintenance Phase | 0 | 0 | 1 | 1 | 0 | 2
  Multiple Races indicated, Maintenance Phase | 0 | 1 | 0 | 0 | 0 | 1
Baseline Serum potassium ( S-K ) levels during both the Acute and Maintenance phases [Number; unit: Participants]
  <5.5 mmol/L, Acute Phase | 119 | 0 | 0 | 0 | 0 | 119
  5.5-<6.0 mmol/L, Acute Phase | 100 | 0 | 0 | 0 | 0 | 100
  ≥ 6.0 mmol/L, Acute Phase | 39 | 0 | 0 | 0 | 0 | 39
  <5.5 mmol/L, Maintenance Phase | 0 | 43 | 23 | 19 | 24 | 109
  5.5-<6.0 mmol/L, Maintenance Phase | 0 | 30 | 17 | 23 | 26 | 96
  ≥ 6.0 mmol/L, Maintenance Phase | 0 | 12 | 5 | 9 | 6 | 32
eGFR at baseline during both the Acute and Maintenance phases [Number; unit: Participants]
  <60 mL/min, Acute Phase | 179 | 0 | 0 | 0 | 0 | 179
  ≥ 60 mL/min, Acute Phase | 72 | 0 | 0 | 0 | 0 | 72
  Not reported, Acute Phase | 7 | 0 | 0 | 0 | 0 | 7
  <60 mL/min, Maintenance Phase | 0 | 52 | 31 | 38 | 41 | 162
  ≥ 60 mL/min, Maintenance Phase | 0 | 28 | 12 | 13 | 15 | 68
  Not reported, Maintenance Phase | 0 | 5 | 2 | 0 | 0 | 7
Etiology of elevated S-K levels during both the Acute and Maintenance phases [Number; unit: Participants] — Categories not mutually exclusive
  Participants
    RAAS inhibitor medication, Acute Phase | 180 | 0 | 0 | 0 | 0 | 180
    Diabetes mellitus, Acute Phase | 170 | 0 | 0 | 0 | 0 | 170
    Chronic kidney disease, Acute Phase | 169 | 0 | 0 | 0 | 0 | 169
    Heart failure, Acute Phase | 94 | 0 | 0 | 0 | 0 | 94
    RAAS inhibitor medication, Maintenance Phase | 0 | 61 | 33 | 36 | 33 | 163
    Diabetes mellitus, Maintenance Phase | 0 | 54 | 26 | 38 | 39 | 157
    Chronic kidney disease, Maintenance Phase | 0 | 50 | 29 | 36 | 37 | 152
    Heart failure, Maintenance Phase | 0 | 26 | 18 | 18 | 25 | 87

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Potassium Between Maintenance Phase Study Days 8 to 29, Inclusive (MP-ITT Population).
Description: The least squares means (LSMeans) are dervied from a mixed effects model of serial log transformed S-K values between Days 8 and 29 with patients as a random effect and the following fixed effects terms: MP treatment group; AP baseline eGFR; AP and MP baseline S-K levels, age categories (<55, 55-64, >= 65 years); and binary indicators for RAAS inhibitors use, CKD, CHF, and DM. The LSmeans estimate obtained from the above model is back-transformed and presented as the lsmeans of all available S-K values during the Maintenance phase study Days 8 to 29.
Time Frame: 22 Days; Maintenance Phase Days 8 - 29, inclusive.
Population: Maintenance Phase Intent- to-Treat (MP-ITT) population: all randomized patients who received at least 1 Maintenance Phase dose and had at least 1 observed S-K assessment on or after Study Day 8.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
mmol/L | 5.0603 [4.9646 to 5.1578] | 4.7544 [4.6350 to 4.8769] | 4.5081 [4.4005 to 4.6184] | 4.3742 [4.2754 to 4.4753]

2. Secondary Outcome: The Number of Normokalemic Days Between Maintenance Phase Study Days 8 to 29, Inclusive (MP-ITT).
Description: The number of normokalemic days during the Maintenance Phase Study Days 8 to 29 is calculated assuming that the interval between assessments is normokalemic only if both the beginning and end assessments for that time interval display normal S-K values (i.e. 3.5 - 5.0 mmol/L)
Time Frame: 22 days; Maintenance Phase Day 8 - 29, inclusive.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
Days | 7.4 (8.0) | 13.4 (7.57) | 13.9 (7.91) | 16.8 (6.99)

3. Secondary Outcome: Mean Change in S-K Levels From Acute Phase Baseline to Maintenance Phase Study Day 2 to Day 29/Exit .
Time Frame: Acute Phase baseline to Maintenance Phase Study Day 2 to Day 29/Exit, inclusive.
Population: Maintenance Phase Intent- to-Treat (MP-ITT) population: all randomized subjects who received at least 1 Maintenance Phase dose and had at least 1 observed S-K assessment on or after Study Day 8.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
mmol/L
  AP Baseline S-K level | 5.55 (0.471) | 5.53 (0.357) | 5.58 (0.423) | 5.55 (0.331)
  MP Study Day 2 Mean Change | -0.86 (0.508) | -1.03 (0.408) | -1.25 (0.471) | -1.12 (0.477)
  MP Study Day 8 Mean Change | -0.49 (0.549) | -0.72 (0.552) | -1.09 (0.629) | -1.20 (0.592)
  MP Study Day 12 Mean Change | -0.41 (0.508) | -0.75 (0.516) | -1.11 (0.663) | -1.20 (0.665)
  MP Study Day 15 Mean Change | -0.48 (0.612) | -0.77 (0.492) | -1.11 (0.652) | -1.19 (0.627)
  MP Study Day 19 Mean Change | -0.45 (0.549) | -0.79 (0.520) | -1.04 (0.581) | -1.07 (0.575)
  MP Study Day 22 Mean Change | -0.45 (0.578) | -0.71 (0.543) | -0.93 (0.653) | -1.05 (0.586)
  MP Study Day 26 Mean Change | -0.43 (0.552) | -0.65 (0.448) | -0.87 (0.697) | -1.03 (0.597)
  MP Study Day 29 Mean Change | -0.47 (0.499) | -0.69 (0.500) | -1.08 (0.704) | -1.12 (0.571)
  MP Study Day 29/Exit Mean Change | -0.44 (0.515) | -0.77 (0.559) | -1.10 (0.813) | -1.19 (0.659)

4. Secondary Outcome: Mean Percent Change in S-K Levels From Acute Phase Baseline to Maintenance Phase Study Day 2 to Day 29/Exit, Inclusive .
Time Frame: Acute Phase baseline to Maintenance Phase Study Day 2 to Day 29/Exit, inclusive.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
Percent Change
  MP Study Day 2 Percent Change | -15.11 (8.154) | -18.53 (6.941) | -22.19 (7.897) | -20.04 (7.959)
  MP Study Day 8 Percent Change | -8.45 (9.492) | -12.84 (9.700) | -19.16 (10.708) | -21.29 (10.135)
  MP Study Day 12 Percent Change | -7.22 (8.967) | -13.36 (8.949) | -19.45 (11.072) | -21.22 (11.368)
  MP Study Day 15 Percent Change | -8.28 (10.739) | -13.73 (8.485) | -19.33 (10.884) | -21.19 (10.675)
  MP Study Day 19 Percent Change | -7.87 (9.554) | -14.08 (8.822) | -18.29 (9.707) | -19.10 (9.957)
  MP Study Day 22 Percent Change | -7.74 (9.992) | -12.65 (9.591) | -16.25 (11.292) | -18.65 (10.034)
  MP Study Day 26 Percent Change | -7.54 (9.386) | -11.83 (8.025) | -15.18 (11.988) | -18.28 (10.271)
  MP Study Day 29 Percent Change | -8.23 (8.586) | -12.49 (8.770) | -18.83 (11.951) | -19.80 (9.503)
  MP Study Day 29/Exit Percent Change | -7.68 (8.940) | -13.85 (9.568) | -19.28 (14.099) | -21.06 (11.086)

5. Secondary Outcome: Mean Change in S-K Levels From Maintenance Phase Baseline to Maintenance Phase Day 2 to Day 29/Exit.
Time Frame: Maintenance phase baseline to Maintenance Phase Study Day 29/Exit, inclusive.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
mmol/L
  MP Baseline S-K level | 4.55 (0.427) | 4.51 (0.357) | 4.38 (0.407) | 4.45 (0.372)
  MP Study Day 2 Mean change | 0.13 (0.411) | -0.01 (0.372) | -0.04 (0.384) | -0.02 (0.400)
  MP Study Day 8 Mean change | 0.50 (0.538) | 0.30 (0.467) | 0.12 (0.523) | -0.10 (0.535)
  MP Study Day 12 Mean change | 0.60 (0.580) | 0.26 (0.541) | 0.10 (0.594) | -0.11 (0.572)
  MP Study Day 15 Mean change | 0.54 (0.694) | 0.25 (0.535) | 0.11 (0.552) | -0.10 (0.546)
  MP Study Day 19 Mean change | 0.55 (0.672) | 0.22 (0.580) | 0.17 (0.483) | 0.01 (0.605)
  MP Study Day 22 Mean change | 0.55 (0.627) | 0.30 (0.563) | 0.27 (0.650) | 0.03 (0.579)
  MP Study Day 26 Mean change | 0.55 (0.623) | 0.34 (0.565) | 0.33 (0.673) | 0.05 (0.594)
  MP Study Day 29 Mean change | 0.52 (0.545) | 0.28 (0.664) | 0.14 (0.668) | -0.04 (0.554)
  MP Study Day 29/Exit Mean change | 0.56 (0.582) | 0.25 (0.645) | 0.11 (0.768) | -0.09 (0.598)

6. Secondary Outcome: Mean Percent Change in S-K Levels From Maintenance Phase Baseline to Maintenance Phase Day 2 to Day 29/Exit.
Time Frame: Maintenance phase baseline to Maintenance Phase Study Day 29/Exit, inclusive.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
Percent Change
  MP Study Day 2 Percent change | 3.39 (9.044) | 0.06 (8.036) | -0.51 (8.862) | -0.20 (8.984)
  MP Study Day 8 Percent change | 11.64 (12.291) | 6.93 (10.486) | 3.05 (12.346) | -1.74 (12.043)
  MP Study Day 12 Percent change | 13.70 (13.072) | 6.38 (12.287) | 2.85 (13.595) | -2.00 (12.836)
  MP Study Day 15 Percent change | 12.51 (15.693) | 5.95 (12.169) | 2.93 (12.662) | -1.89 (12.118)
  MP Study Day 19 Percent change | 12.96 (15.791) | 5.33 (12.934) | 4.28 (11.231) | .095 (13.697)
  MP Study Day 22 Percent change | 12.84 (14.342) | 6.98 (12.774) | 6.79 (15.174) | 1.39 (12.782)
  MP Study Day 26 Percent change | 13.03 (14.566) | 7.98 (12.932) | 8.08 (15.516) | 1.88 (16.641)
  MP Study Day 29 Percent change | 12.09 (13.116) | 6.12 (14.424) | 3.02 (17.785) | -1.43 (13.664)
  MP Study Day 29/Exit Percent change | 12.97 (13.116) | 6.12 (14.424) | 3.02 (17.785) | -1.43 (13.664)

7. Secondary Outcome: Median Time to Hyperkalemia (S-K ≥ 5.1mmol/L)
Time Frame: Maintenance Phase baseline to maintenance Phase Study Day 29/Exit.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
Days | 7 [6 to 7] | 14 [7 to 28] | NA [NA to NA] — The Median time was not reached in the ZS 10 g group because fewer than 50% of patients in the group had a hyperkalemic event before the end of the Maintenance Phase. | NA [NA to NA] — The Median time was not reached in the ZS 15 g group because fewer than 50% of patients in the group had a hyperkalemic event before the end of the Maintenance Phase.

8. Secondary Outcome: Mean S-K Intra-subject Standard Deviation Calculated Among Subjects With ≥ 2 Values on or After Maintenance Phase Study Day 8
Time Frame: 22 days; Maintenance Phase Day 8 - 29
Population: Maintenance Phase Intent- to-Treat (ITT) population: all randomized subjects who received at least 1 Maintenance Phase dose and had at least 1 observed S-K assessment on or after Day 8.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
mmol/L | 0.06392 [0.05804 to 0.06980] | 0.06367 [0.05574 to 0.07159] | 0.07708 [0.06941 to 0.08474] | 0.06849 [0.06126 to 0.07571]

9. Secondary Outcome: Proportion of Subjects Who Remained Normokalemic During Maintenance Phase
Time Frame: Maintenance Phase Study Days 1, 2, 5, 8, 12, 15, 19, 22, 26, 29, and 35, inclusive.
Population: as for outcome 3
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
Proportion of subjects
  Baseline | 0.866 | 0.933 | 0.920 | 0.926
  MP Study Day 2 | 0.84 | 0.933 | 0.918 | 0.944
  MP Study Day 8 | 0.481 | 0.711 | 0.820 | 0.852
  MP Study Day 12 | 0.400 | 0.750 | 0.787 | 0.849
  MP Study Day 15 | 0.438 | 0.705 | 0.851 | 0.827
  MP Study Day 19 | 0.449 | 0.744 | 0.787 | 0.882
  MP Study Day 22 | 0.442 | 0.674 | 0.667 | 0.882
  MP Study Day 26 | 0.486 | 0.738 | 0.711 | 0.843
  MP Study Day 29 | 0.507 | 0.667 | 0.816 | 0.907
  MP Study Day 29/Exit | 0.476 | 0.711 | 0.760 | 0.852

10. Secondary Outcome: Median Time to Relapse in S-K Values
Description: Median time to relapse in S-K values (return to original Acute Phase S-K baseline value)
Time Frame: Maintenance phase Study Day 1 to Study Day 29/Exit.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Number analyzed (Participants) | 82 | 45 | 50 | 54
Days | 19 [12 to 28] | 29 [29 to NA] — The confidence interval for the median is based on when the lower and upper limits of the confidence interval for survival function reach 50%. However, the upper limit for survival function in the ZS 5 g QD did not reach 50% in the Maintenance Phase. | NA [NA to NA] — Fewer than 50% of patients in the ZS 10 g QD had relapsed at the end of the Maintenance Phase. Therefore, median was not reached. | NA [NA to NA] — Fewer than 50% of patients in the ZS 15 g QD had relapsed at the end of the Maintenance Phase. Therefore, median was not reached.

11. Secondary Outcome: Exponential Rate of Change in S-K Values During the Acute Phase at 24 Hours and 48 Hours of Study Drug Treatment.
Time Frame: Acute Phase 24 hours and Acute Phase 48 hours.
Population: Acute Phase ITT Population included all subjects who received at least 1 Acute Phase dose and had any post-baseline S-K levels after receiving the investigational product during the first 48 hours.
Measure: Mean (Standard Error); unit: log(mmol/L/hour)
Groups:
- Acute Phase: ZS 10 g TID: ZS (sodium zirconium cyclosilicate) 10 g, three times a day, orally as suspension in water for 48 hours.
Arm/Group | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 258
log(mmol/L/hour)
  24 hours after start of ZS dosing | -0.00373 (0.000231)
  48 hours of start of ZS dosing | -0.00324 (0.000130)

12. Secondary Outcome: Mean Change From Baseline in S-K Values (Blood) at All Measured Time Intervals Post Dose Acute Phase.
Time Frame: All measured time intervals post dose during the Acute Phase.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 258
mmol/L
  Acute phase baseline | 5.55 (0.449)
  1 hour after start of ZS dosing Mean change | -0.23 (0.435)
  2 hours after start of ZS dosing Mean change | -0.41 (0.440)
  4 hours after start of ZS dosing Mean change | -0.51 (0.405)
  24 hours after start of ZS dosing Mean change | -0.68 (0.448)
  1 hour after 1st dose Study Day 2 Mean change | -0.75 (0.444)
  48 hours after start of ZS dosing Mean change | -1.05 (0.510)

13. Secondary Outcome: Mean Percent Change From Baseline in S-K Values (Blood) at All Measured Time Intervals Post Dose Acute Phase.
Time Frame: All measured time intervals post dose during the Acute Phase.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 258
Percent Change
  1 hour after start of ZS dosing Percent change | -3.91 (7.741)
  2 hours after start of ZS dosing Percent change | -7.13 (7.706)
  4 hours after start of ZS dosing Percent change | -9.00 (7.123)
  24 hours after start of ZS dosing Percent change | -12.03 (7.808)
  1 hour after 1st dose Study Day 2 Percent change | -13.41 (7.720)
  48 hours after start of ZS dosing Percent change | -18.56 (8.506)

14. Secondary Outcome: Proportion of Subjects Who Achieve Normokalemia During the Acute Phase at 24 and 48 Hours After Start of Dosing
Time Frame: Through 48 hours acute phase
Population: as for outcome 11
Measure: Number; unit: Proportion of subjects
Arm/Group | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 258
Proportion of subjects
  24 hours after start of dosing | 0.661
  48 hours after of start dosing | 0.88

15. Secondary Outcome: Median Time to Normalization (3.50-5.0 mmol/L) in S-K Levels in the 48 Hours of Initial Treatment
Time Frame: Through 48 hours acute phase
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Hours
Groups:
- Acute Phase: ZS 10 g TID: ZS (sodium zirconium cyclosilicate) 10 g, three times a day, orally as a suspension for 48 hours.
Arm/Group | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 258
Hours | 2.17 [2 to 3.97]

ADVERSE EVENTS:
Time Frame: All adverse events were collected beginning with the first administration of study drug and through end of study treatment follow up visit. End of treatment study follow up visit was 7 days +/- 1 day after last dose of investigational product.
Groups:
- ZS 10 g TID (Acute Phase): ZS (sodium zirconium cyclosilicate) 10 g, three times a day, orally as suspension in water for 48 hours.
Arm/Group | ZS 10 g TID (Acute Phase) | Placebo Comparator (Maintenance Phase) | ZS 5 g Once Daily (Maintenance Phase) | ZS 10 g Once Daily (Maintenance Phase) | ZS 15 g Once Daily (Maintenance Phase)
Serious Adverse Events (participants affected / at risk) | 0/258 | 0/85 | 5/45 | 2/51 | 3/56
Other Adverse Events (participants affected / at risk) | 9/258 | 25/85 | 20/45 | 15/51 | 25/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZS 10 g TID (Acute Phase) (N=258) | Placebo Comparator (Maintenance Phase) (N=85) | ZS 5 g Once Daily (Maintenance Phase) (N=45) | ZS 10 g Once Daily (Maintenance Phase) (N=51) | ZS 15 g Once Daily (Maintenance Phase) (N=56)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Generalized edema (General disorders) | 0 | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZS 10 g TID (Acute Phase) (N=258) | Placebo Comparator (Maintenance Phase) (N=85) | ZS 5 g Once Daily (Maintenance Phase) (N=45) | ZS 10 g Once Daily (Maintenance Phase) (N=51) | ZS 15 g Once Daily (Maintenance Phase) (N=56)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 6 | 0 | 1 | 1
Edema (General disorders) | 0 | 2 | 1 | 3 | 8 — Including generalized and peripheral edema
Fatigue (General disorders) | 0 | 0 | 0 | 5 | 6
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Upper respiratory infection (Infections and infestations) | 1 | 1 | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Dysponea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Generalised Oedema (General disorders) | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 2 | 0 | 3 | 6
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZS Pharma has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.